CLINICAL TRIAL: NCT01987037
Title: Neuropsychomotor Functions in Children With Autism Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Bertrand Olliac, M.D Ph.D., Centre Hospitalier Esquirol
Other Study IDs: 2013-A00644-41
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; neuropsychomotor assessment; NP-MOT; motor skills; gross motor
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tests evaluation: children with autism spectrum disorder subjected to the NP-MOT tests
  Interventions: Behavioral: neuropsychomotor assessment

INTERVENTIONS:
Behavioral: neuropsychomotor assessment — Children with autism spectrum disorders pass a specific battery test (NP-MOT) for a neuropsychomotor assessment. This neuropsychomotor assessment is administered in a half-day maximum. This battery aims to investigate passive muscle tone (shoulders, limbs, and trunk), standing and synkinesia, static and dynamic balance, tonic laterality (extensibility and dangling of hands and feet to identify the tonic dominant side), laterality of use, fine-digit movements, digital tactile gnosis, and body spatial integration (knowing left from right: for oneself and that of others, and with regard to objects).

SUMMARY:
The aim of the study is to describe the feasibility of the passation of the assessment battery of psychomotor functions tests (NP-MOT) in children aged 4 to 11 years with a diagnosis of autism spectrum disorder: number and type of evaluable events, number and type of tests with a deficit compared to the standard results.

DETAILED DESCRIPTION:
After informed consent obtention, the children will be submitted to the different tests of the battery to evaluate the psychomotor functions. The results will be compared with other data collected from the routine practise : socio-demographic data, medical and developmental antecedents,psychological tests (KABC II, Rey test, London Tower test, ...), psychomotor evaluation (MABC, evaluation of manual praxis, visual abilities, Frostig test), understanding data (N-EEL test), neuropediatric examination, clinical assessment (ADI-R, CARS).

The use of this battery allows this fine discriminative assessment of the psychomotor functions involved in the movement. Exploring each function will allow to take into account qualitative and quantitative aspects of the movement in every aspects, and this is not applied in the routine care until now. Calibration for each event can explore each function independently of each other, and will provide information to determine any specific developmental characteristics improve care.

ELIGIBILITY:
Inclusion Criteria:

* informed consent from the parents or the legal representative
* age 4 to 11
* autism spectrum disorder diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition- text revised

Exclusion Criteria:

* bad understanding of the french language
* motor disability from lesion or accidental origin, proved genetic or neurologic disease
* deafness, blindness
* parents with administrative or judiciary protection, and without health insurance

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children attended in the Centre Hospitalier Esquirol and the CRA (Autism Reference Center) in Limousin, France, for suspiscion of autism
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
results to the NP-MOT tests battery | one day
  the NP-MOT battery tests include several tests to evaluate 9 motor functions (muscle tone, gross motor, laterality, fine-digit movement, digital tactile gnosis, hand-eye skill, body spatial orientation, pace, auditory attention) with 48 subtests.
  We describe:
  number and type of evaluable tests, number and type of tests with results with 1 Standard Deviation different from the standard results.
  number and type of tests with results with 2 Standard Deviation different from the standard results.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de Ressources Autisme Limousin, Limoges
  - Centre Hospitalier esquirol, Limoges

REFERENCES:
- [Background] Lasserre E, Vaivre-Douret L, Abadie V. Psychomotor and cognitive impairments of children with CHARGE syndrome: common and variable features. Child Neuropsychol. 2013 Sep;19(5):449-65. doi: 10.1080/09297049.2012.690372. Epub 2012 Jun 14. PMID 23906312